CLINICAL TRIAL: NCT00569621
Title: A Randomized, Double-Masked, Placebo-Controlled Two Cross Over Study Comparing the Effects of Moxaverine and Placebo on Ocular Blood Flow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dorothea Gross, Ursapharm Arzneimittel GmbH & Co. KG
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOXOPH1
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia | interventions — moxaverine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Moxaverine
- 2 (Placebo Comparator)
  Interventions: Drug: physiological saline

INTERVENTIONS:
Drug: Moxaverine — intravenous administration
  Arms: 1
Drug: physiological saline — intravenous administration
  Arms: 2

SUMMARY:
It is known that several common eye diseases are associated with ocular perfusion abnormalities. Moxaverine is used in the therapy of perfusion abnormalities in the brain, the heart and the extremities because of its direct vasodilatory effects. The present study seeked to investigate whether moxaverine alters ocular blood flow in healthy volunteers after intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

* 6 healthy volunteers of either sex
* Age 18-35 yrs.
* Body mass index between 15th and 85th percentile, nonsmokers

Exclusion Criteria:

* Regular use of medication
* Abuse of alcoholic beverages or drugs
* Participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Ametropy less 3 dpt
* Acute gastric bleeding, massive cerebral hemorrhage related to stroke
* Women: pregnancy or lactation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Retinal and Choroidal Blood flow | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, Prof, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria